CLINICAL TRIAL: NCT02667886
Title: A Phase 1/2 Trial of X4P-001 as Single Agent and in Combination With Axitinib in Patients With Advanced Renal Cell Carcinoma
Brief Title: Trial of X4P-001 in Participants With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-RCCA
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Results first posted 2024-08-14 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — mavorixafor; Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Part A): X4P-001 200 mg BID with Axitinib (Experimental): Participants will receive X4P-001 200 milligrams (mg) orally twice daily (BID) with axitinib at 5 mg orally BID.
  Interventions: Drug: X4P-001; Drug: axitinib
- Dose Escalation (Part A): X4P-001 400 mg QD with Axitinib (Experimental): Participants will receive X4P-001 400 mg orally once daily (QD) with axitinib at 5 mg orally BID.
  Interventions: Drug: X4P-001; Drug: axitinib
- Dose Escalation (Part A): X4P-001 600 mg QD with Axitinib (Experimental): Participants will receive X4P-001 600 mg orally QD with axitinib at 5 mg orally BID.
  Interventions: Drug: X4P-001; Drug: axitinib
- Dose Expansion (Part B): X4P-001 400 mg QD With Axitinib (Experimental): Participants received X4P-001 400 mg orally QD with axitinib at 5 mg orally BID.
  Interventions: Drug: X4P-001; Drug: axitinib
- Dose Escalation and Expansion (Part C): X4P-001 600 mg QD Monotherapy (Experimental): Participants will receive X4P-001 600 mg orally QD.
  Interventions: Drug: X4P-001

INTERVENTIONS:
Drug: X4P-001 — Continuous, oral dosing
  Other Names: Mavorixafor; AMD11070
Drug: axitinib — Continuous, oral dosing
  Other Names: Inlyta
  Arms: Dose Escalation (Part A): X4P-001 200 mg BID with Axitinib; Dose Escalation (Part A): X4P-001 400 mg QD with Axitinib; Dose Escalation (Part A): X4P-001 600 mg QD with Axitinib; Dose Expansion (Part B): X4P-001 400 mg QD With Axitinib

SUMMARY:
The purpose of the study is to test different doses of X4P-001 given alone and in combination with axitinib in participants diagnosed with advanced renal cell carcinoma. The goals of the study are to determine the safety and tolerability of X4P-001, as well as the potential effect it may have on the body and the cancer tumor.

DETAILED DESCRIPTION:
X4P-001 is an orally bioavailable C-X-C chemokine receptor type 4 (CXCR4) antagonist that has demonstrated activity in various tumor models. CXCR4 is the receptor for C-X-C chemokine ligand type 12 (CXCL12). CXCL12 has potent chemotactic activity for lymphocytes and myeloid-derived suppressor cells (MDSCs), and is important in homing of hematopoietic stem cells to the bone marrow. CXCR4 is also expressed and active on multiple types of human cancers, including clear cell Renal Cell Carcinoma (ccRCC), ovarian cancer, and melanoma, and increased expression of CXCR4 on tumor cells has been associated with significantly decreased overall participant survival.

Multiple observations implicate the CXCL12/CXCR4 axis in contributing to the lack (or loss) of tumor responsiveness to angiogenesis inhibitors (also referred to as "angiogenic escape"). In animal cancer models, interference with CXCR4 function has been demonstrated to disrupt the tumor microenvironment and unmask the tumor to immune attack by multiple mechanisms, including:

* Eliminating tumor re-vascularization
* Decreasing the infiltration of MDSCs
* Increasing the ratio of cluster of differentiation 8+ (CD8+) T cells to T regulatory (Treg) cells

The hypothesis and evidence of published data support is that effective CXCR4 antagonism by X4P-001 would be of potential benefit in participants with advanced ccRCC and other cancers by multiple mechanisms:

* Decreased recruitment of MDSCs, resulting in increased anti-tumor immune attack
* Sustained decrease in neoangiogenesis and tumor vascular supply
* Interference with the autocrine effect of increased expression by ccRCC of both CXCR4 and CXCL12, its only ligand, thereby, potentially reducing cancer cell metastasis

This initial clinical trial in participants with advanced ccRCC will evaluate X4P-001 both as a single agent (monotherapy) and also in combination with axitinib, a small molecule tyrosine kinase inhibitor (TKI) approved for second-line treatment of participants with ccRCC. This combination has the potential to further improve outcomes by reducing the angiogenic escape that typically occurs with TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of predominant ccRCC.
* Have received at least one prior course of treatment for ccRCC. Part C only: Prior treatment must include at least 1 course of vascular endothelial growth factor (VEGF)-directed therapy.
* Have on computed tomography (CT) imaging done within 28 days of Day 1 findings consistent with advanced ccRCC, including at least one extra-renal measurable target lesion meeting the criteria of Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
* For women of childbearing potential and men, agree to use effective contraceptive methods from screening, through the study, and for at least 4 weeks after the last dose of study drug.
* For women of childbearing potential, have a negative pregnancy test (serum or urine) on Day 1 prior to initiating study treatment.
* Be willing and able to comply with the protocol

Exclusion Criteria:

* Has life expectancy of less than 3 months.
* Has performance status Grade >2 (Eastern Cooperative Oncology Group [ECOG] criteria).
* Has New York Heart Association (NYHA) Class III or IV heart failure or uncontrolled hypertension (systolic blood pressure [SBP] ≥160 millimeters of mercury [mm Hg]; diastolic blood pressure [DBP] ≥100 mm Hg).
* Has previously received X4P-001.
* Parts A and B only: Has received a prior course of axitinib.
* Parts A and B only: Has received mechanistic target of rapamycin (mTOR) inhibitor(s) as their only prior treatment for ccRCC.
* Has a prior history or current evidence of intracranial (CNS) metastatic RCC, except for

  ≤3 lesions treated by CyberKnife or excisional surgery, clinically stable for at least 4 weeks, and without evidence of recurrence on MRI imaging at screening.
* Has ongoing acute clinical adverse events National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade >1 resulting from prior cancer therapies (except alopecia, tyrosine kinase inhibitor [TKI]-related hand-foot syndrome, or thyroid dysfunction).
* Has had within the past 6 months the occurrence or persistence of one or more of the following medical conditions that could not be controlled with usual medical care (for example, required emergency care or hospitalization): hypertension, angina, congestive heart failure, diabetes, seizure disorder.
* Has had within the past 6 months the occurrence of one or more of the following events: myocardial infarction, cerebrovascular accident, deep vein thrombosis, pulmonary embolism, hemorrhage (CTC Grade 3 or 4), chronic liver disease (meeting criteria for Child-Pugh Class B or C), a second active malignancy (excluding basal cell carcinoma and cervical carcinoma in situ), organ transplantation.
* Has had within the 4 weeks prior to initiation of study drug, or is expected to have during the study period, surgery requiring general anesthesia.
* Has, at screening, serologic laboratory tests meeting one or more of the following criteria:
* An indeterminate or positive test for antibody to human immunodeficiency virus (HIV)-1 or -2.
* An indeterminate or positive test for antibody to hepatitis C virus (HCV), unless documented to have no detectable viral load on two independent samples.
* A positive test for hepatitis B surface antigen (HBsAg).
* Has, at screening, safety laboratory tests meeting one or more of the following criteria:
* Hemoglobin <8.0 grams (g)/deciliter (dL)
* Absolute neutrophil count (ANC) <1,500/microliter (μL)
* Platelets <75,000/μL
* Creatinine >2.0x upper limit of normal (ULN)
* Serum aspartate transaminase (AST) >2.5x ULN
* Serum alanine transaminase (ALT) >2.5x ULN
* Total bilirubin >1.5x ULN (unless due to Gilbert's Syndrome)
* International normalized ratio (INR) >1.5x ULN
* Has received other anti-cancer therapy within the following specified intervals prior to Day 1:
* TKI within 2 weeks.
* Radiation therapy within 2 weeks.
* Bevacizumab within 4 weeks.
* Other chemotherapy (for example, mitomycin-C, nitrosourea) or immunotherapy (for example, antibody, cytokine) within 4 weeks
* For investigational anti-cancer therapies, the interval will be determined in consultation with the Medical Monitor.
* Has, within 2 weeks prior to Day 1, received a medication prohibited based on cytochrome P3A4 (CYP3A4) interaction
* Has, within 2 weeks prior to Day 1, received systemic corticosteroids exceeding prednisone 10 mg per day or equivalent; for other immunosuppressive agents, the exclusionary dose and duration will be determined in consultation with the Medical Monitor.
* Is, within 2 weeks prior to Day 1, nursing.
* Has, at the planned initiation of study drug, an uncontrolled infection.
* Has any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the participant, or may preclude the participant's successful completion of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-04-27 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (18):
  - Scottsdale, Arizona
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Hackensack, New Jersey
  - New York, New York
  - The Bronx, New York
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - Greenville, South Carolina
  - Houston, Texas
- South Korea (2):
  - Gyeyang-gu, Seoul
  - Seongdu, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study comprised 3 parts: Part A (Phase 1: Dose escalation cohorts), Part B (Phase 2: Dose expansion cohort), and Part C (Dose escalation and expansion cohort). As planned, the efficacy and safety data collected per dose level not per study part.
Groups:
- Dose Escalation (Part A): X4P-001 200 mg BID With Axitinib: Participants received X4P-001 200 milligrams (mg) orally twice daily (BID) with axitinib at 5 mg orally BID.
- Dose Escalation (Part A): X4P-001 400 mg QD With Axitinib: Participants received X4P-001 400 mg orally once daily (QD) with axitinib at 5 mg orally BID.
- Dose Escalation (Part A): X4P-001 600 mg QD With Axitinib: Participants received X4P-001 600 mg orally QD with axitinib at 5 mg orally BID.
- Dose Escalation and Expansion (Part C): X4P-001 600 mg QD Monotherapy: Participants received X4P-001 600 mg orally QD.
Period: Dose Escalation (Part A)
Arm/Group | Dose Escalation (Part A): X4P-001 200 mg BID With Axitinib | Dose Escalation (Part A): X4P-001 400 mg QD With Axitinib | Dose Escalation (Part A): X4P-001 600 mg QD With Axitinib | Dose Expansion (Part B): X4P-001 400 mg QD With Axitinib | Dose Escalation and Expansion (Part C): X4P-001 600 mg QD Monotherapy
Started | 3 | 7 | 6 | 0 | 0
Received at Least 1 Dose of Study Drug | 3 | 7 | 6 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0
Not Completed | 2 | 7 | 6 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 0 | 0
Not completed — Disease Progression | 1 | 4 | 3 | 0 | 0
Not completed — Dose-limiting toxicity (DLT) | 0 | 0 | 2 | 0 | 0
Period: Dose Expansion (Part B)
Arm/Group | Dose Escalation (Part A): X4P-001 200 mg BID With Axitinib | Dose Escalation (Part A): X4P-001 400 mg QD With Axitinib | Dose Escalation (Part A): X4P-001 600 mg QD With Axitinib | Dose Expansion (Part B): X4P-001 400 mg QD With Axitinib | Dose Escalation and Expansion (Part C): X4P-001 600 mg QD Monotherapy
Started | 0 | 0 | 0 | 55 | 0
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 55 | 0
Completed | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 54 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 9 | 0
Not completed — Clinical Deterioration | 0 | 0 | 0 | 3 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 38 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 0
Period: Dose Escalation and Expansion (Part C)
Arm/Group | Dose Escalation (Part A): X4P-001 200 mg BID With Axitinib | Dose Escalation (Part A): X4P-001 400 mg QD With Axitinib | Dose Escalation (Part A): X4P-001 600 mg QD With Axitinib | Dose Expansion (Part B): X4P-001 400 mg QD With Axitinib | Dose Escalation and Expansion (Part C): X4P-001 600 mg QD Monotherapy
Started | 0 | 0 | 0 | 0 | 3
Received at Least 1 Dose of Study Drug | 0 | 0 | 0 | 0 | 3
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — DLT | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug. As planned, Baseline Characteristics data collected per dose level not per study part.
Groups:
- X4P-001 200 mg BID With Axitinib: Participants received X4P-001 200 mg orally BID with axitinib at 5 mg orally BID in Part A.
- X4P-001 400 mg QD With Axitinib: Participants received X4P-001 400 mg orally QD with axitinib at 5 mg orally BID in either Part A or Part B.
- X4P-001 600 mg QD With Axitinib: Participants received X4P-001 600 mg orally QD with axitinib at 5 mg orally BID in Part A.
- X4P-001 600 mg QD Monotherapy: Participants received X4P-001 600 mg orally QD in Part C.
- Total: Total of all reporting groups
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib | X4P-001 600 mg QD With Axitinib | X4P-001 600 mg QD Monotherapy | Total
Number analyzed (Participants) | 3 | 62 | 6 | 3 | 74
Age, Customized [Count of Participants; unit: Participants]
  16-64 Years | 3 | 37 | 4 | 1 | 45
  ≥65 Years | 0 | 25 | 2 | 2 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 10 | 0 | 2 | 12
  Male | 3 | 52 | 6 | 1 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 7 | 0 | 0 | 7
  Not Hispanic or Latino | 3 | 55 | 6 | 3 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 17 | 0 | 0 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 2
  White | 3 | 40 | 6 | 3 | 52
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Parts A, B, and C: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An SAE was an AE that met at least 1 of the following criteria: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization for the AE, persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), important medical event or reaction. Adverse events with onset after administration of the first dose of study drug up to 10 days after last dosing date were considered TEAEs. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: From first dose of study drug up to 10 days after last dosing (maximum exposure: 52.1 months)
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib | X4P-001 600 mg QD With Axitinib | X4P-001 600 mg QD Monotherapy
Number analyzed (Participants) | 3 | 62 | 6 | 3
Participants | 3 | 62 | 6 | 3

2. Secondary Outcome: Parts A and B: Objective Response Rate (ORR), as Assessed Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: The ORR was defined as percentage of participants with best overall response of complete response (CR) or partial response (PR). CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to <10 millimeters (mm). PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From administration of first dose of study medication until disease progression, study completion or early termination (up to 80 weeks)
Population: Clinically evaluable population included all participants who received at least 1 dose of study medication, who had at least 1 valid post-baseline response (CR/PR/stable disease [SD]/progressive disease [PD]) and had no major protocol deviations which impacted the efficacy assessment. Due to dose-limiting toxicities (DLTs) experienced by participants, the sample size was too small for data to be collected for this Outcome Measure for the "X4P-001 600 mg QD With Axitinib" arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib
Number analyzed (Participants) | 3 | 59
percentage of participants | 66.7 [9.4 to 99.2] | 27.1 [16.4 to 40.3]

3. Secondary Outcome: Parts A and B: Time to Objective Response, as Assessed Using RECIST v1.1
Description: Time to objective response was defined as time from first administration of combination regimen to first CR or PR whichever came first. CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From administration of first dose of study medication until first appearance of CR or PR (up to 80 weeks)
Population: Clinically evaluable population included all participants who received at least 1 dose of study medication, who had at least 1 valid post-baseline response (CR/PR/SD/PD) and had no major protocol deviations which impacted the efficacy assessment. Due to DLTs experienced by participants, the sample size was too small for data to be collected for this Outcome Measure for the "X4P-001 600 mg QD With Axitinib" arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib
Number analyzed (Participants) | 3 | 59
months | 12.9 [1.9 to NA] — Due to smaller number of participants with an event, upper limit of 95% confidence interval (CI) could not be calculated. | 14.6 [12.9 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated.

4. Secondary Outcome: Parts A and B: Duration of Objective Response (DOR), as Assessed Using RECIST v1.1
Description: The DOR was defined as the time from first CR or PR whichever came first until the time of disease progression or death by any cause. CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Disease progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of 1 or more new lesions was also considered progression.
Time Frame: Time from first CR or PR until the time of disease progression or death due to any cause (up to 80 weeks)
Population: Clinically evaluable population included all participants who received at least 1 dose of study medication, who had at least 1 valid post-baseline response (CR/PR/SD/PD) and had no major protocol deviations which impacted efficacy assessment. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. Due to DLTs experienced by participants, the sample size was too small for data to be collected for this Outcome Measure for "X4P-001 600 mg QD With Axitinib" arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib
Number analyzed (Participants) | 2 | 16
months | NA [9.2 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated. | 16.6 [10.8 to 36.0]

5. Secondary Outcome: Parts A and B: Disease Control Rate (DCR), as Assessed Using RECIST v1.1
Description: The DCR was defined as the percentage of participants with best overall response of CR, PR or stable disease (SD). CR: Disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) with a reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. The appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib
Number analyzed (Participants) | 3 | 59
percentage of participants | 100.0 [29.2 to 100.0] | 71.2 [57.9 to 82.2]

6. Secondary Outcome: Parts A and B: Time to Progression (TTP), as Assessed Using RECIST v1.1
Description: The TTP was defined as the time from first administration of combination regimen until PD. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions or the appearance of 1 or more new lesions was also considered progression.
Time Frame: From administration of first dose of study medication until disease progression (up to 80 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib
Number analyzed (Participants) | 3 | 59
months | 11.1 [5.5 to NA] — Due to smaller number of participants with an event, upper limit of 95% CI could not be calculated. | 7.4 [5.6 to 14.7]

7. Secondary Outcome: Parts A and B: Progression Free Survival (PFS), as Assessed Using RECIST v1.1
Description: The PFS was defined as the time from first administration of combination regimen until disease progression or death from any cause. Disease progression: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum also demonstrated an absolute increase of at least 5 mm. An unequivocal progression of existing non-target lesions or the appearance of 1 or more new lesions was also considered progression.
Time Frame: From administration of first dose of study medication until disease progression or death from any cause (up to 80 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib
Number analyzed (Participants) | 3 | 59
months | 11.1 [5.5 to NA] — Due to smaller number of participants with an event, the upper limit of 95% CI could not be calculated. | 7.4 [5.5 to 12.5]

8. Secondary Outcome: Parts A and B: Maximum Plasma Concentration (Cmax) of X4P-001
Time Frame: Day 1 and Day 15 of Cycle 1
Population: The pharmacokinetic (PK) population included all participants who had at least one evaluable concentration. Here 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms (ng)/milliliter (mL)
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib | X4P-001 600 mg QD With Axitinib
Number analyzed (Participants) | 3 | 57 | 6
nanograms (ng)/milliliter (mL)
  Day 1 | 1070 (59.5) | 3130 (67.2) | 4170 (42.7)
  Day 15: number analyzed (Participants) | 2 | 53 | 5
  Day 15 | 831 (8.20) | 3710 (73.5) | 3900 (39.2)

9. Secondary Outcome: Area Under the Curve From Time 0 to the Last Quantifiable Timepoint (AUC0-tlast)
Time Frame: Day 1 and Day 15 of Cycle 1
Population: The PK population included all participants who had at least one evaluable concentration. Here 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib | X4P-001 600 mg QD With Axitinib
Number analyzed (Participants) | 3 | 57 | 6
hours*ng/mL
  Day 1 | 2200 (62.8) | 6790 (80.2) | 9830 (54.3)
  Day 15: number analyzed (Participants) | 2 | 53 | 5
  Day 15 | 3000 (26.4) | 13100 (90.7) | 15100 (44.3)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 10 days after last dosing (maximum exposure: 52.1 months)
Description: Safety population included all participants who received at least 1 dose of study drug. As planned, safety data collected per dose level not per study part.
Arm/Group | X4P-001 200 mg BID With Axitinib | X4P-001 400 mg QD With Axitinib | X4P-001 600 mg QD With Axitinib | X4P-001 600 mg QD Monotherapy
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/62 | 1/6 | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 26/62 | 1/6 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 62/62 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | X4P-001 200 mg BID With Axitinib (N=3) | X4P-001 400 mg QD With Axitinib (N=62) | X4P-001 600 mg QD With Axitinib (N=6) | X4P-001 600 mg QD Monotherapy (N=3)
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acquired tracheooesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cholestatic liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Device failure (Product Issues) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | X4P-001 200 mg BID With Axitinib (N=3) | X4P-001 400 mg QD With Axitinib (N=62) | X4P-001 600 mg QD With Axitinib (N=6) | X4P-001 600 mg QD Monotherapy (N=3)
Diarrhoea (Gastrointestinal disorders) | 3 | 33 | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 22 | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 20 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 12 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 11 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 9 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 8 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 4 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 5 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 5 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral papule (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 28 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 16 | 3 | 1
Alanine aminotransferase increased (Investigations) | 0 | 8 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 7 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 4 | 1 | 0
Lipase increased (Investigations) | 1 | 3 | 1 | 0
White blood cell count increased (Investigations) | 0 | 4 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 3 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 3 | 0 | 0
Weight increased (Investigations) | 0 | 3 | 0 | 1
Amylase increased (Investigations) | 0 | 2 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0 | 0
Blood fibrinogen increased (Investigations) | 0 | 2 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 2 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 2 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Tri-iodothyronine decreased (Investigations) | 0 | 1 | 0 | 0
Thyroid function test abnormal (Investigations) | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0
Blood albumin increased (Investigations) | 0 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0
Vitamin d decreased (Investigations) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 30 | 5 | 2
Chills (General disorders) | 0 | 8 | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 6 | 0 | 0
Influenza like illness (General disorders) | 0 | 6 | 0 | 0
Pyrexia (General disorders) | 0 | 6 | 0 | 0
Asthenia (General disorders) | 1 | 3 | 1 | 0
Oedema peripheral (General disorders) | 0 | 5 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 4 | 0 | 0
Chest pain (General disorders) | 0 | 4 | 0 | 0
Gait disturbance (General disorders) | 1 | 3 | 0 | 0
Pain (General disorders) | 0 | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 1 | 0
Facial pain (General disorders) | 0 | 2 | 0 | 0
Decreased activity (General disorders) | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0
Suprapubic pain (General disorders) | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 32 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 10 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 6 | 3 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 3 | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 16 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 14 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 12 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 12 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 9 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 9 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 13 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 8 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 4 | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 2 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 3 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 24 | 3 | 0
Hot flush (Vascular disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 2 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 10 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 7 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 10 | 2 | 0
Vision blurred (Eye disorders) | 1 | 5 | 0 | 1
Eye pain (Eye disorders) | 0 | 2 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 2 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 1 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 1 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0
Macular oedema (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinal pigmentation (Eye disorders) | 0 | 1 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment 0 (Eye disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 6 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Dermatophytosis of nail (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Pyuria (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 4 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 4 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 3 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 14 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 12 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 6 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 1 | 0
Depression (Psychiatric disorders) | 0 | 3 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 3 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 1 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 6 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0/0 | 1/10 | 0/0 | 0/2 — This is a sex-specific AE. Only female participants were at risk.
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1/52 | 0 | 0/1 — This is a sex-specific AE. Only male participants were at risk.
Gynaecomastia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1/52 | 0 | 0/1 — This is a sex-specific AE. Only male participants were at risk.
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0/0 | 1/10 | 0/0 | 0/2 — This is a sex-specific AE. Only female participants were at risk.
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hepatobiliary disorders (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic vascular thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0 | 0
Electrocardiogram Q wave abnormal (Investigations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Localised Oedema (General disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/86/NCT02667886/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT02667886/SAP_001.pdf